CLINICAL TRIAL: NCT02236806
Title: Role of ACE Inhibitors and Beta Blockers as Cardiotoxicity Prevention in Breast Cancer Patients Treated With (Neo)Adjuvant Anthracyclines and/or Trastuzumab: a Four Arm, Placebo Control, Randomized Trial
Brief Title: Cardiotoxicity Prevention in Breast Cancer Patients Treated With Anthracyclines and/or Trastuzumab
Acronym: SAFE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SAFE2014
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Cardiotoxicity
Keywords: Breast cancer; Adjuvant chemotherapy; Neoadjuvant chemotherapy; Cardioprotection; Anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Bisoprolol; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both participants and Care Providers are not aware of intervention allocation.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): bisoprolol plus ramipril
  Interventions: Drug: Bisoprolol; Drug: Ramipril
- Arm 2 (Active Comparator): Bisoprolol plus placebo
  Interventions: Drug: Bisoprolol; Drug: Placebo
- Arm 3 (Active Comparator): Ramipril plus placebo
  Interventions: Drug: Ramipril; Drug: Placebo
- Arm 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — 5 mg daily
  Arms: Arm 1; Arm 2
Drug: Ramipril — 5 mg daily
  Arms: Arm 1; Arm 3
Drug: Placebo — 1 capsule daily
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
The aim of the study is to analyze the protective impact on the cardiac damage of beta blockers and ACE inhibitors for breast cancer patients treated with anthracyclines-based chemotherapy with or without trastuzumab.

DETAILED DESCRIPTION:
Over the years, due to the use of new generation therapeutic regimens, as well as the use of advanced radiation techniques, the curability of breast cancer reached an overall 10-year survival rate of approximately 80%.

Anthracyclines have a key role in the treatment of breast cancer. Many published studies showed a benefit of disease-free survival in patients with positive lymph nodes treated with anthracyclines-based regimens. Many anthracyclines and taxanes-based regimens are currently used in clinical practice in the treatment of breast cancer. Numerous randomized trials have confirmed the benefit of the addition of taxanes to anthracyclines.

Trastuzumab is a recombinant humanized monoclonal antibody with specificity for the extracellular domain of human epidermal growth factor receptor 2 (HER2). The use of trastuzumab administered sequentially or concurrently with adjuvant chemotherapy compared to chemotherapy in patients with HER2 positive was evaluated in several randomized trials. Many data concerning the incidence of adverse cardiovascular events acute, subacute and late are now available. The cardiac toxicity of anthracyclines may be acute, subacute and chronic. The acute toxicity occurs during or shortly after the infusion of the drug with arrhythmias, which in some cases leads to heart failure, pericarditis-myocarditis and electrocardiographic abnormalities. The acute toxicity is usually reversible in a dose-dependent manner. The acute and subacute toxicity are rare (1-4%). Data are available concerning clinically relevant cardiac toxicity with a chronic progressive deterioration of ventricular function up to heart failure.

Beside the cumulative dose risk factor, other unfavourable features such as advanced age, female sex, and the combination of anthracyclines and trastuzumab should be evaluated. In most cases, the late toxicity occurs within the first year following completion of chemotherapy but nevertheless the clinical manifestations can occur even after 10-20 years. This fact suggests that in women treated in (neo)adjuvant setting is strongly necessary an echocardiographic monitoring even after a longer time.

The aim of the study is to analyze the protective impact on the cardiac damage of beta blockers and ACE inhibitors for breast cancer patients treated with anthracyclines-based chemotherapy with or without trastuzumab, using myocardial strain imaging monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age >18 years
* Non-metastatic histologically confirmed primary invasive breast cancer
* Scheduled to receive neoadjuvant and/or adjuvant anthracyclines with or without anti-HER2 therapy
* Provided informed consent
* Able to swallow capsules
* LVEF > 50%

Exclusion Criteria:

* Pregnant or lactating women
* Treatment with ACE-inhibitors or beta blockers at diagnosis
* History of NCI Common Toxicity Criteria for Adverse Effects (CTCAE) (version 4.0) Grade >2 symptomatic congestive heart failure (CHF), previous myocardial infarction, significant symptoms (Grade>2) relating to LVEF dysfunction, valvular disease, cardiac arrhythmia (Grade>3)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | at months 6,9,12,24
  Change in LVEF (3-dimensional and 2-dimensional) at time-frame
Global longitudinal strain (GLS) | at months 6,9,12,24
  Change in GLS at time-frame

SECONDARY OUTCOMES:
Indexed left ventricular end diastolic volume (EDVI) | at months 6,9,12,24
  Change in EDVI at time-frame
Indexed left ventricular end systolic volume (ESVI) | at months 6,9,12,24
  Change in ESVI at time-frame

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, MD, Prof, Study Chair — Azienda Ospedaliero-Universitaria Careggi; Icro Meattini, MD, Prof, Principal Investigator — University of Florence
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi, Florence University, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francolini G, Desideri I, Meattini I, Becherini C, Terziani F, Olmetto E, Delli Paoli C, Pezzulla D, Loi M, Bonomo P, Greto D, Calusi S, Casati M, Pallotta S, Livi L. Assessment of a guideline-based heart substructures delineation in left-sided breast cancer patients undergoing adjuvant radiotherapy : Quality assessment within a randomized phase III trial testing a cardioprotective treatment strategy (SAFE-2014). Strahlenther Onkol. 2019 Jan;195(1):43-51. doi: 10.1007/s00066-018-1388-x. Epub 2018 Nov 7. PMID 30406290
- [Background] Meattini I, Curigliano G, Terziani F, Becherini C, Airoldi M, Allegrini G, Amoroso D, Barni S, Bengala C, Guarneri V, Marchetti P, Martella F, Piovano P, Vannini A, Desideri I, Tarquini R, Galanti G, Barletta G, Livi L. SAFE trial: an ongoing randomized clinical study to assess the role of cardiotoxicity prevention in breast cancer patients treated with anthracyclines with or without trastuzumab. Med Oncol. 2017 May;34(5):75. doi: 10.1007/s12032-017-0938-x. Epub 2017 Mar 31. PMID 28364270
- [Result] Livi L, Barletta G, Martella F, Saieva C, Desideri I, Bacci C, Del Bene MR, Airoldi M, Amoroso D, Coltelli L, Scotti V, Becherini C, Visani L, Salvestrini V, Mariotti M, Pedani F, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Olivotto I, Meattini I. Cardioprotective Strategy for Patients With Nonmetastatic Breast Cancer Who Are Receiving an Anthracycline-Based Chemotherapy: A Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1544-1549. doi: 10.1001/jamaoncol.2021.3395. PMID 34436523
- [Derived] Marrazzo L, Meattini I, Becherini C, Salvestrini V, Visani L, Barletta G, Saieva C, Del Bene MR, Pilato G, Desideri I, Arilli C, Paoletti L, Russo S, Scoccianti S, Martella F, Francolini G, Simontacchi G, Nori Cucchiari J, Pellegrini R, Livi L, Pallotta S. Subclinical cardiac damage monitoring in breast cancer patients treated with an anthracycline-based chemotherapy receiving left-sided breast radiation therapy: subgroup analysis from a phase 3 trial. Radiol Med. 2024 Dec;129(12):1926-1935. doi: 10.1007/s11547-024-01897-6. Epub 2024 Oct 22. PMID 39436588